CLINICAL TRIAL: NCT03232944
Title: Personalized CRT - Multiple Point Pacing Post Approval Study
Brief Title: Personalized CRT - MPP Post Approval Study
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: MPP PAS
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- CRT non-responders with MPP enabled: Patients enrolled and implanted with a CRT Quad system, who are identified as CRT non-responder, for which MPP is enabled.
  Interventions: Device: Cardiac Resynchronization Therapy - MPP

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy - MPP — The multiple point pacing feature (MPP) is designed to allow pacing from 2 LV electrodes.

SUMMARY:
The purpose of this Post-Approval Study (PAS) is to evaluate the effectiveness of MPP to improve CRT response in the non-responder patient population when used in "real-world" clinical practice, following commercial release. This evaluation is based on the Clinical Composite Score which summarizes the proportions and frequencies of CRT non-responder patients who are "improved", "unchanged" or "worsened" after receiving MPP therapy. Patients will be followed for the duration of the PAS. This study is required by FDA as a condition of approval of the MPP feature and is integrated within the Product Surveillance Registry (PSR).

DETAILED DESCRIPTION:
Medtronic market-released cardiac resynchronization therapy (CRT) Quadripolar (Quad) systems approved for commercial release with the Multiple Point Pacing (MPP) feature were eligible to contribute to the Post-Approval Study (PAS) objectives. Products with MPP capabilities receiving appropriate license or regulatory approval during the conduct of the PAS were included and contributed to the PAS objectives upon commercial release. CRT is an established pacing therapy for patients with heart failure (HF). CRT provides atrial- synchronized biventricular (BiV) pacing using standard pacing technology combined with a special third lead that is implanted via the coronary sinus and positioned in a cardiac vein to sense and/or pace the left ventricle (LV). Following a sensed atrial contraction or atrial paced event, both ventricles are stimulated to synchronize their contraction. The MPP feature is designed to allow a second LV pace to occur in LV Only or BiV pace configurations. In the LV Only pace configuration, the LV paces occur simultaneously or sequentially (LV- LV), as applicable by product. When Bi-V pacing is enabled, the RV pace can be delivered either before or after the LV paces, with the order determined by the programmed Ventricular Pacing Configuration.

The MPP PAS was a global, prospective, observational multi-center study. Patients implanted with an eligible CRT Quad system were enrolled and followed in the Product Surveillance Registry per the expected standard of care practices of their care provider.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient has or is intended to receive or be treated with an eligible CRT device
* Patient within 30 days of therapy received at the time of their initial PSR platform enrollment

Exclusion Criteria:

* Patient who is, or is expected to be inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes patients that are or will be implanted with an eligible CRT Quad system.
Sampling Method: Non-Probability Sample
Enrollment: 1338 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
MPP therapy responder | Up to 3 years
  To estimate the proportion of MPP therapy responders among patients who did not respond to standard CRT and had MPP programmed "on".

SECONDARY OUTCOMES:
HF hospitalization and/or mortality | Up to 3 years
  Summarize incidence of HF hospitalization and/or mortality probability after MPP enabled

CONTACTS AND LOCATIONS:
Locations (78):
- United States (46):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Saint Vincent Heart Clinic Arkansas, Little Rock, Arkansas
  - Chula Vista Cardiac Center, Chula Vista, California
  - Desert Heart Rhythm Consultants, Palm Springs, California
  - COR Healthcare, Torrance, California
  - Colorado Springs Cardiology, Colorado Springs, Colorado
  - Denver Heart, Denver, Colorado
  - Colorado Heart and Vascular, PC, Lakewood, Colorado
  - Heart Rhythm Solutions, Hollywood, Florida
  - Baptist Health, Jacksonville, Florida
  - Heart & Vascular Institute of Florida, Safety Harbor, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - The University of Kansas Medical Center, Kansas City, Kansas
  - MedStar Health Research Institute, Baltimore, Maryland
  - The Johns Hopkins Hospital, Bethesda, Maryland
  - Delmarva Heart Research Foundation Inc, Salisbury, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - UP Health System - Marquette, Marquette, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - North Memorial Heart and Vascular Institute, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Missouri Cardiovascular Specialists, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - HealthCare Partners Medical Group, Henderson, Nevada
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - Island Cardiac Specialists, Garden City, New York
  - Huntington Hospital, Huntington, New York
  - Northwell Health, Manhasset, New York
  - Hudson Valley Heart Center, Poughkeepsie, New York
  - Central New York Cardiology, Utica, New York
  - WakeMed Health & Hospitals, Raleigh, North Carolina
  - Northeast Ohio Cardiovascular Specialists, Akron, Ohio
  - The Christ Hospital Health Network, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Mercy Health - Saint Vincent Medical Center, Toledo, Ohio
  - Cleveland Clinic, Cleveland, Oklahoma
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Saint Thomas Research Institute, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - Kootenai Heart Clinics Northwest, Spokane, Washington
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin
- Belgium (2):
  - UZ Leuven - Campus Gasthuisberg, Leuven
  - CHU UCL Mont-Godinne - Dinant, Yvoir
- Canada (2):
  - Montreal Heart Institute, Montreal, Quebec
  - Institut de cardiologie et de pneumologie de Québec (IUCPQ), Québec, Quebec
- France (6):
  - CHRU Brest - Hôpital de la Cavale Blanche, Brest
  - Centre Hospitalier Universitaire de Clermont-Ferrand - Gabriel-Montpied, Clermont-Ferrand
  - CHRU La Rochelle, La Rochelle
  - CHU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - Nouvelles Cliniques Nantaises, Nantes
  - Centre hospitalier de la région d'Annecy, Pringy
- Germany (6):
  - Universitätsklinikum Aachen, AöR, Aachen
  - St. Vinzenz-Hospital Köln, Cologne
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum des Saarlandes, Homburg
  - Eberhard Karls Universität Tübingen - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Magyar Honvédség Honvédkorház, Budapest, Hungary
- Azienda Ospedaliera Ospedale Niguarda Cà Granda, Milan, Italy
- Institut Jantung Negara - National Heart Institute, Kuala Lumpur, Malaysia
- Netherlands (2):
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Maasstad Hospital Rotterdam, Rotterdam
- Vychodoslovensky ustav srdcovych a cievnych chorob, a.s., Košice, Slovakia
- Samsung Medical Center, Seoul, South Korea
- Spain (4):
  - Hospital Universitario da Coruña, A Coruña
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela
- United Kingdom (5):
  - University Hospitals of Birmingham NHS Foundation Trust - Queen Elizabeth Hospital, Birmingham
  - Glenfield Hospital, Leicester
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - Central Manchester University Hospitals NHS - Manchester Royal Infirmary, Manchester
  - The James Cook University Hospital - South Tees Hospitals NHS, Middlesbrough